CLINICAL TRIAL: NCT02341625
Title: A Phase I/IIa Study of BMS-986148, a Mesothelin Directed Antibody Drug Conjugate, in Subjects With Select Advanced Solid Tumors
Brief Title: A Study of BMS-986148 in Patients With Select Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study terminated for business reasons not related to safety.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA008-002; 2014-002485-70 (EudraCT Number)
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: Ascending dose of BMS-986148 (Experimental): BMS-986148 Intravenous injection at increasing doses on specific days until the maximum tolerated dose is reached. Five cancers will be studied in this part: mesothelioma, pancreatic, ovarian, gastric, and non-small cell lung cancer. Alternate dose and schedules may be explored.
  Interventions: Drug: BMS-986148
- Part 2: Expansion dose of BMS-986148 (Experimental): BMS-986148 Intravenous injection of Maximum tolerated dose (MTD) on specific days. Five cancers will be studied in this part: mesothelioma, pancreatic, ovarian, gastric, and non-small cell lung cancer.
  Interventions: Drug: BMS-986148
- Part 3A: Ascending dose of BMS-986148 (Experimental): Set dose of nivolumab and BMS-986148 intravenous injection at increasing doses on specific days until the maximum tolerated dose is reached. Five cancers will be studied in this part: mesothelioma, pancreatic, ovarian, gastric, and non-small cell lung cancer.
  Interventions: Drug: BMS-986148; Biological: Nivolumab
- Part 3B: Expansion dose of BMS-986148 (Experimental): Set dose of nivolumab and BMS-986148 intravenous injection at or below maximum tolerated dose on specific days. Five cancers will be studied in this part: mesothelioma, pancreatic, ovarian, gastric, and non-small cell lung cancer.
  Interventions: Drug: BMS-986148; Biological: Nivolumab

INTERVENTIONS:
Drug: BMS-986148
Biological: Nivolumab
  Other Names: Opdivo
  Arms: Part 3A: Ascending dose of BMS-986148; Part 3B: Expansion dose of BMS-986148

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics, immunogenicity, antitumor activity and pharmacodynamics of BMS-986148 administered alone and in combination with nivolumab in patients with mesothelioma, non-small cell lung cancer, ovarian cancer, pancreatic cancer and gastric cancer.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have pancreatic, ovarian, gastric, non-small cell cancer or mesothelioma. For dose expansion, must have tumor that is positive for mesothelin
* Expected to have life expectancy of at least 3 months
* Men and women 18 years old or older (or local age of majority)
* Must have measurable tumor per Response Evaluation Criteria In Solid Tumors (RECIST) or modified RECIST for malignant pleural mesothelioma
* ECOG of 0 to 1

Exclusion Criteria:

* Cancer metastases in the brain
* Moderate eye disorders
* Active infection or past hepatitis B or C infection
* Major surgery less than 1 month before the start of the study
* Uncontrolled heart disease
* Impaired liver or bone marrow function
* History of allergy to mesothelin-directed antibodies, tubulysin, monoclonal antibodies, nivolumab or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-06-19 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2020-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (2):
  - Moores Cancer Center, La Jolla, California
  - Duke University Medical Center, Durham, North Carolina
- Australia (4):
  - Local Institution - 0013, Liverpool, New South Wales
  - Local Institution - 0014, Adelaide, South Australia
  - Local Institution - 0004, Clayton, Victoria
  - Local Institution - 0015, Nedlands, Western Australia
- Belgium (2):
  - Local Institution - 0008, Ghent, Oost-Vlaanderen
  - Local Institution - 0009, Brussels
- Canada (2):
  - Local Institution - 0002, Edmonton, Alberta
  - Local Institution - 0003, Toronto, Ontario
- Italy (3):
  - Local Institution - 0017, Milan, Lombardy
  - Local Institution - 0018, Milan
  - Local Institution - 0016, Rozzano (milano)
- Netherlands (2):
  - Local Institution - 0010, Amsterdam
  - Local Institution - 0011, Rotterdam
- United Kingdom (2):
  - Local Institution - 0007, Southampton, Hampshire
  - Local Institution - 0006, Glasgow, Lanarkshire

REFERENCES:
- [Derived] Rottey S, Clarke J, Aung K, Machiels JP, Markman B, Heinhuis KM, Millward M, Lolkema M, Patel SP, de Souza P, Duca M, Curigliano G, Santoro A, Koyama T, Brown M, Vezina H, He C, Chu QS. Phase I/IIa Trial of BMS-986148, an Anti-mesothelin Antibody-drug Conjugate, Alone or in Combination with Nivolumab in Patients with Advanced Solid Tumors. Clin Cancer Res. 2022 Jan 1;28(1):95-105. doi: 10.1158/1078-0432.CCR-21-1181. Epub 2021 Oct 6. PMID 34615718
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- BMS-986148 0.1MG/KG Q3W: Part 1A Dose Escalation: BMS-986148 0.1 mg/kg IV Q3W in a 21-day cycle
- BMS-986148 0.2MG/KG Q3W: Part 1A Dose Escalation: BMS-986148 0.2 mg/kg IV Q3W in a 21-day cycle
- BMS-986148 0.4MG/KG Q3W: Part 1A Dose Escalation: BMS-986148 0.4 mg/kg IV Q3W in a 21-day cycle
- BMS-986148 0.8MG/KG Q3W: Part 1A Dose Escalation: BMS-986148 0.8 mg/kg IV Q3W in a 21-day cycle
- BMS-986148 1.2MG/KG Q3W Es: Part 1A Dose Escalation BMS-986148 1.2 mg/kg IV Q3W
- BMS-986148 1.6MG/KG Q3W: Part 1A Dose Escalation: BMS-986148 1.6 mg/kg IV Q3W in a 21-day cycle
- BMS-986148 1.2MG/KG Q3W Ex: Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
- BMS-986148 0.4MG/KG QW: Part 1B Dose Escalation: BMS-986148 0.4 mg/kg IV QW for 3 weeks and 1 week off in a 28-day cycle
- BMS-986148 0.6MG/KG QW: Part 1B Dose Escalation: BMS-986148 0.6 mg/kg IV QW for 3 weeks and 1 week off in a 28-day cycle
- BMS-986148 0.8MG/KG Q3W+Nivolumab: Part 3A Dose Escalation: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W in a 21-day cycle
  Part 3B Dose Expansion: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
Period: Overall Study
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab
Started | 2 | 2 | 3 | 8 | 8 | 10 | 51 | 8 | 4 | 30
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 3 | 8 | 8 | 10 | 51 | 8 | 4 | 30
Not completed — Disease Progression | 2 | 2 | 3 | 6 | 7 | 7 | 28 | 5 | 4 | 19
Not completed — Study Drug Toxicity | 0 | 0 | 0 | 1 | 0 | 3 | 10 | 0 | 0 | 3
Not completed — Adverse Event Unrelated to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Not completed — Participant Request to Discontinue Study Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 2 | 0 | 0
Not completed — Participant Withdrew Consent | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Completed Treatment as per Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other Reasons | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 2
Not completed — Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- BMS 0.8MG/KG + Nivolumab Q3W: Part 3A Dose Escalation: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W in a 21-day cycle
  Part 3B Dose Expansion: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
- Total: Total of all reporting groups
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG + Nivolumab Q3W | Total
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 8 | 10 | 51 | 8 | 4 | 30 | 126
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.5 (0.7) | 70.5 (0.7) | 65.3 (5.8) | 63.9 (5.4) | 63.4 (5.1) | 59.0 (16.0) | 61.5 (9.5) | 66.3 (8.6) | 64.5 (9.1) | 61.6 (9.4) | 62.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 2 | 3 | 3 | 3 | 31 | 3 | 2 | 12 | 59
  Male | 2 | 2 | 1 | 5 | 5 | 7 | 20 | 5 | 2 | 18 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3 | 8 | 8 | 10 | 46 | 8 | 3 | 25 | 114
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 1 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3
  White | 1 | 2 | 3 | 7 | 7 | 9 | 46 | 8 | 3 | 30 | 116
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events at Worst CTC Grade
Description: Number of participants with adverse events at worst CTC grade including any grade adverse events (AEs), serious adverse events (SAEs), adverse events leading to discontinuations, and deaths grouped by dose + dose regimen.
Time Frame: From first dose to up to 100 days post last dose (Up to 6 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Groups:
- BMS-986148 1.2MG/KG Q3W Es: Part 1A Dose Escalation BMS-986148 1.2 mg/kg IV Q3W
  Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 59 | 8 | 4 | 30
Participants
  Adverse Events (AEs) | 1 | 2 | 3 | 8 | 10 | 59 | 8 | 4 | 30
  Serious Adverse Events (SAEs) | 1 | 1 | 1 | 5 | 4 | 32 | 6 | 3 | 21
  AEs Leading to Discontinuation | 0 | 0 | 0 | 1 | 3 | 11 | 1 | 0 | 7
  Deaths | 1 | 2 | 3 | 5 | 7 | 38 | 7 | 4 | 22

2. Primary Outcome: Number of Participants With Laboratory Test Toxicity Grade Shifting From Baseline
Description: Number of participants with laboratory test toxicity grade (Grade 0, 1, 2, 3, and 4) in hematology and chemistry shifting from baseline. An increase in baseline indicates a shift of participant to a greater toxicity grade. A decrease in baseline indicates a shift of participant to a lesser toxicity grade. Participants are grouped by dose + dose regimen assessed by NCT CTCAE V 4.03.
Time Frame: From first dose to up to 100 days post last dose (Up to 6 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 59 | 8 | 4 | 30
Participants
  Hemoglobin increase from baseline | 1 | 1 | 0 | 3 | 3 | 20 | 2 | 1 | 12
  Hemoglobin decrease from baseline | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0
  Platelet Count increase from baseline | 0 | 0 | 0 | 3 | 4 | 14 | 0 | 1 | 6
  Platelet Count decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes increase from baseline | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 2
  Leukocytes decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Neutrophils increase from baseline | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1
  Neutrophils decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Lymphocytes increase from baseline | 1 | 2 | 1 | 3 | 6 | 27 | 6 | 3 | 19
  Lymphocytes decrease from baseline | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Absolute Neutrophil increase from baseline | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 2
  Absolute Neutrophil decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Alkaline Phosphatase (ALP) increase from baseline | 0 | 1 | 1 | 6 | 10 | 46 | 5 | 4 | 24
  Alkaline Phosphatase (ALP) decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (AST) increase from baseline | 0 | 1 | 1 | 6 | 10 | 53 | 6 | 4 | 26
  Aspartate Aminotransferase (AST) decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase (ALT) increase from baseline | 0 | 0 | 0 | 7 | 10 | 50 | 5 | 3 | 25
  Alanine Aminotransferase (ALT) decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Bilirubin increase from baseline | 0 | 1 | 0 | 2 | 3 | 16 | 2 | 2 | 7
  Bilirubin decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine increase from baseline | 0 | 0 | 1 | 2 | 2 | 7 | 1 | 3 | 5
  Creatinine decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium increase from baseline | 0 | 1 | 1 | 4 | 4 | 23 | 1 | 2 | 17
  Sodium decrease from baseline | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium increase from baseline | 1 | 0 | 0 | 3 | 5 | 24 | 1 | 2 | 9
  Potassium decrease from baseline | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
  Calcium Total increase from baseline | 0 | 0 | 0 | 5 | 4 | 17 | 3 | 1 | 10
  Calcium Total decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Calcium Corrected increase from baseline | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
  Calcium Corrected decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Phosphorus increase from baseline | 2 | 0 | 2 | 3 | 4 | 24 | 1 | 2 | 7
  Phosphorus decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Magnesium increase from baseline | 0 | 1 | 1 | 2 | 4 | 22 | 1 | 2 | 5
  Magnesium decrease from baseline | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
  Glucose Fasting Serum increase from baseline | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 5
  Glucose Fasting Serum decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Albumin increase from baseline | 0 | 1 | 0 | 7 | 8 | 37 | 6 | 2 | 19
  Albumin decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Amylase increase from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Amylase decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase increase from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Lipase decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatine Kinase increase from baseline | 0 | 0 | 1 | 0 | 0 | 9 | 0 | 0 | 3
  Creatine Kinase decrease from baseline | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Uric Acid increase from baseline | 0 | 0 | 1 | 1 | 2 | 6 | 0 | 2 | 6
  Uric Acid decrease from baseline | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Maximum observed serum concentration (Cmax) of BMS-986148 grouped by dose + dose regimen.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: PK blood assessed on cycle 1, day 1
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Groups:
- BMS 1.2MG/KG Q3W Ex: Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
- BMS 0.8MG/KG Q3W+Nivolumab Es: Part 3A Dose Escalation: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W in a 21-day cycle
- BMS 0.8MG/KG Q3W+Nivolumab Ex: Part 3B Dose Expansion: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG Q3W+Nivolumab Es | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 8 | 49 | 8 | 4 | 11 | 17
ug/mL
  Total Antibody: number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Total Antibody | 2.3 (31.4) | 2.8 (7.6) | 3.3 (76.7) | 16.4 (47.2) | 39.8 (24.5) | 28.5 (14.0) | 28.3 (22.5) | 9.3 (21.3) | 14.5 (22.3) | 16.7 (19.7) | 18.8 (22.4)
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Active Antibody-Drug Conjugate (ADC) | 2.0 (29.8) | 2.2 (8.2) | 2.6 (76.1) | 15.8 (46.4) | 40.0 (26.3) | 27.0 (18.6) | 27.5 (22.6) | 8.8 (20.3) | 13.6 (31.0) | 15.3 (27.6) | 17.8 (24.6)
  Unconjugated Tubulysin: number analyzed (Participants) | 0 | 0 | 1 | 4 | 9 | 8 | 45 | 2 | 2 | 5 | 11
  Unconjugated Tubulysin |  |  | 0.5 (NA) — Too few events to calculate arithmetic coefficient of variation | 0.2 (17.1) | 0.4 (52.3) | 0.4 (70.9) | 0.3 (58.2) | 0.1 (36.0) | 0.4 (75.0) | 0.2 (42.5) | 0.2 (42.5)

4. Secondary Outcome: Time of Maximum Observed Serum Concentration (Tmax)
Description: Time of maximum observed serum concentration (Tmax) of BMS-986148 grouped by dose + dose regimen.
Time Frame: PK blood assessed on cycle 1, day 1
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG Q3W+Nivolumab Es | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 8 | 49 | 8 | 4 | 11 | 17
Hours
  Total Antibody: number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Total Antibody | 2.2 [0.3 to 4.0] | 2.2 [0.3 to 4.1] | 3.9 [0.5 to 4.7] | 4.0 [0.2 to 4.8] | 3.9 [0.9 to 4.3] | 4.1 [1.1 to 4.1] | 4.0 [0.8 to 24.1] | 4.0 [0.6 to 4.1] | 3.8 [1.1 to 3.9] | 1.1 [0.6 to 24.1] | 4.0 [0.9 to 23.8]
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Active Antibody-Drug Conjugate (ADC) | 0.2 [0.1 to 0.3] | 2.2 [0.3 to 4.1] | 0.5 [0.1 to 3.9] | 2.5 [0.2 to 4.0] | 1.5 [0.8 to 4.3] | 3.8 [1.0 to 4.1] | 3.9 [0.8 to 4.7] | 4.0 [0.6 to 4.1] | 3.8 [1.1 to 3.9] | 1.0 [0.6 to 4.2] | 4.0 [0.9 to 4.0]
  Unconjugated Tubulysin: number analyzed (Participants) | 0 | 0 | 1 | 4 | 9 | 8 | 45 | 2 | 2 | 5 | 11
  Unconjugated Tubulysin |  |  | 25.5 [25.5 to 25.5] | 120.2 [71.8 to 169.7] | 167.3 [71.4 to 170.0] | 168.8 [48.0 to 335.5] | 166.1 [24.3 to 338.8] | 168.2 [166.9 to 169.4] | 166.7 [94.7 to 238.7] | 165.1 [48.0 to 170.9] | 166.5 [47.8 to 335.9]

5. Secondary Outcome: Concentration at the End of a Dosing Interval (Ctau)
Description: Concentration at the end of a dosing interval (Ctau) of BMS-986148 grouped by dose + dose regimen.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: PK blood assessed on cycle 1, day 1
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG Q3W+Nivolumab Es | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 2 | 8 | 10 | 7 | 46 | 8 | 3 | 10 | 17
ug/mL
  Total Antibody: number analyzed (Participants) | 2 | 2 | 2 | 8 | 8 | 7 | 46 | 8 | 3 | 9 | 17
  Total Antibody | 0.0035 (112.0) | 0.0333 (115.7) | 0.8233 (131.8) | 0.4426 (106.1) | 1.4101 (101.8) | 1.0917 (91.9) | 1.1938 (98.7) | 3.2035 (20.2) | 3.8872 (46.1) | 0.2133 (114.0) | 0.7544 (83.5)
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 0 | 1 | 8 | 10 | 7 | 46 | 8 | 3 | 10 | 17
  Active Antibody-Drug Conjugate (ADC) | 0.0633 (141.3) |  | 0.0058 (NA) — Too few events to calculate arithmetic coefficient of variation | 0.0309 (123.8) | 0.3049 (110.0) | 0.2121 (111.3) | 0.1558 (123.4) | 1.2705 (39.5) | 1.9068 (59.1) | 0.1119 (187.1) | 0.0797 (103.7)
  Unconjugated Tubulysin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 2 | 2 | 0 | 1
  Unconjugated Tubulysin |  |  |  |  | 0.1630 (0.9) | 0.2590 (77.1) | 0.1634 (48.2) | 0.1388 (36.0) | 0.3539 (75.0) |  | 0.1330 (NA) — Too few events to calculate arithmetic coefficient of variation

6. Secondary Outcome: Trough Observed Serum Concentration (Ctrough)
Description: Trough observed serum concentration (Ctrough) of BMS-986148 grouped by dose + dose regimen.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: PK blood assessment include cycle 2-day 1 and cycle 1-day 8
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG Q3W+Nivolumab Es | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 3 | 7 | 6 | 8 | 39 | 8 | 3 | 10 | 13
ug/mL
  Total Antibody: number analyzed (Participants) | 2 | 2 | 3 | 7 | 6 | 8 | 38 | 8 | 3 | 10 | 12
  Total Antibody | 0.1 (0.0) | 0.1 (0.00) | 0.1 (0.00) | 0.79676 (92.4) | 0.92146 (125.9) | 1.23291 (81.7) | 1.14568 (104.4) | 3.20352 (20.2) | 3.88717 (46.1) | 0.33875 (122.1) | 0.77912 (79.1)
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 2 | 3 | 7 | 6 | 8 | 38 | 8 | 3 | 10 | 12
  Active Antibody-Drug Conjugate (ADC) | 0.1 (0.0) | 0.1 (0.00) | 0.1 (0.00) | 0.27671 (95.3) | 0.21835 (152.7) | 0.36894 (90.7) | 0.31524 (111.4) | 1.27047 (39.5) | 1.90678 (59.1) | 0.18096 (97.4) | 0.24389 (81.0)
  Unconjugated Tubulysin | 0.00005 (0.0) | 0.00005 (0.0) | 0.00005 (0.0) | 0.00005 (0.0) | 0.00007 (66.6) | 0.00009 (127.6) | 0.00006 (80.7) | 0.00006 (64.7) | 0.00018 (104.0) | 0.00005 (0.0) | 0.00005 (40.8)

7. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Time T (AUC(0-t))
Description: Area under the concentration-time curve from time Zero to time T (AUC(0-t)) of BMS-986148 grouped by dose + dose regimen.
  Note: The geometric CV was not calculated. Arithmetic % CV is reported instead.
Time Frame: PK blood assessment include cycle 1-day 1
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 8 | 51 | 8 | 4 | 11 | 19
h*ug/mL
  Total Antibody: number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Total Antibody | 152.6 (31.6) | 232.5 (17.5) | 129.6 (131.3) | 1979.5 (69.6) | 5399.8 (40.1) | 4285.7 (29.3) | 3472.6 (47.1) | 858.0 (22.9) | 1278.8 (35.1) | 1815.8 (43.4) | 2611.3 (33.5)
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 7 | 49 | 8 | 4 | 11 | 17
  Active Antibody-Drug Conjugate (ADC) | 88.6 (48.7) | 70.7 (42.9) | 60.8 (136.2) | 1042.1 (68.6) | 3083.6 (32.3) | 2493.1 (25.1) | 1984.7 (45.7) | 565.4 (30.3) | 927.3 (38.7) | 1059.0 (44.8) | 1447.5 (36.2)
  Unconjugated Tubulysin: number analyzed (Participants) | 0 | 0 | 1 | 4 | 9 | 8 | 45 | 2 | 2 | 5 | 11
  Unconjugated Tubulysin |  |  | 49.6 (NA) — Too few events to calculate arithmetic coefficient of variation | 29.6 (42.8) | 80.1 (73.4) | 197.0 (59.4) | 42.3 (80.4) | 9.3 (73.0) | 42.5 (84.3) | 25.5 (58.8) | 17.7 (110.3)

8. Secondary Outcome: Area Under the Concentration-Time Curve in One Dosing Interval (AUC[TAU])
Description: Area under the concentration-time curve in one dosing interval (AUC[TAU]) of BMS-986148 grouped by dose + dose regimen Note: The geometric CV was not calculated. Arithmetic % CV is reported instead
Time Frame: PK blood assessment include cycle 1-day 1
Population: All participants who received at least one dose of BMS-986148 and have evaluable serum concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS 0.8MG/KG Q3W+Nivolumab Es | BMS 0.8MG/KG Q3W+Nivolumab Ex
Number analyzed (Participants) | 2 | 2 | 2 | 8 | 10 | 7 | 46 | 8 | 3 | 10 | 17
h*ug/mL
  Total Antibody: number analyzed (Participants) | 2 | 2 | 2 | 8 | 8 | 7 | 46 | 8 | 3 | 9 | 17
  Total Antibody | 179.3 (34.8) | 265.7 (13.3) | 344.6 (98.5) | 2059.3 (68.7) | 5318.6 (36.9) | 4316.1 (28.8) | 4159.4 (39.5) | 858.0 (22.9) | 1533.5 (19.2) | 1839.0 (45.4) | 2689.9 (34.0)
  Active Antibody-Drug Conjugate (ADC): number analyzed (Participants) | 2 | 0 | 1 | 8 | 10 | 7 | 46 | 8 | 3 | 10 | 17
  Active Antibody-Drug Conjugate (ADC) | 109.0 (35.2) |  | 371.6 (NA) — Too few events to calculate arithmetic coefficient of variation | 1098.7 (67.5) | 3246.0 (36.6) | 2507.2 (24.7) | 2271.7 (40.1) | 565.4 (30.3) | 1063.9 (32.2) | 1094.9 (48.0) | 1478.1 (36.6)
  Unconjugated Tubulysin: number analyzed (Participants) | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 2 | 2 | 0 | 1
  Unconjugated Tubulysin |  |  |  |  | 173.4 (48.2) | 197.0 (59.4) | 148.9 (30.3) | 9.3 (73.0) | 42.5 (84.3) |  | 102.4 (NA) — Too few events to calculate arithmetic coefficient of variation

9. Secondary Outcome: Best Overall Response (BOR)
Description: Best overall response is defined as the best response designation over the study as a whole, recorded between the dates of first dose until the last tumor assessment prior to subsequent therapy.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 58 months
Population: Per-protocol, data for this Outcome Measure was collected by disease irrespective of dose. All treated participants are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung Cancer (NSCLC), and Gastric)
Measure: Count of Participants; unit: Participants
Groups:
- BMS-986148 Mesothelioma; BMS-986148 Ovarian: Part 1A Dose Escalation: BMS-986148 starting with a dose of 0.1 mg/kg IV Q3W to a dose of 1.6 mg/kg IV Q3W in a 21-day cycle
  Part 1B Dose Escalation: BMS-986148 starting with a dose of 0.4 mg/kg IV QW to a dose of 0.6 mg/kg IV QW for 3 weeks and 1 week off in a 28-day cycle
  Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
- BMS-986148+Nivolumab Mesothelioma; BMS-986148+Nivolumab Ovarian; BMS-986148+Nivolumab Pancreatic; BMS-986148+Nivolumab NSCLC; BMS-986148+Nivolumab Gastric: Part 3A Dose Escalation: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W in a 21-day cycle
  Part 3B Dose Expansion: BMS-986148 0.8 mg/kg IV Q3W + Nivolumab 360 mg Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
- BMS-986148 Pancreatic; BMS-986148 NSCLC; BMS-986148 Gastric: Part 1A Dose Escalation: BMS-986148 starting with a dose of 0.8 mg/kg IV Q3W to a dose of 1.6 mg/kg IV Q3W in a 21-day cycle
  Part 1B Dose Escalation: BMS-986148 starting with a dose of 0.4 mg/kg IV QW to a dose of 0.6 mg/kg IV QW for 3 weeks and 1 week off in a 28-day cycle
  Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer.
Arm/Group | BMS-986148 Mesothelioma | BMS-986148+Nivolumab Mesothelioma | BMS-986148 Ovarian | BMS-986148+Nivolumab Ovarian | BMS-986148 Pancreatic | BMS-986148+Nivolumab Pancreatic | BMS-986148 NSCLC | BMS-986148+Nivolumab NSCLC | BMS-986148 Gastric | BMS-986148+Nivolumab Gastric
Number analyzed (Participants) | 25 | 13 | 22 | 2 | 18 | 6 | 4 | 2 | 3 | 1
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 13 | 8 | 11 | 2 | 4 | 1 | 1 | 1 | 1 | 0
  Progressive Disease (PD) | 7 | 1 | 7 | 0 | 11 | 2 | 2 | 1 | 2 | 1

10. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate is defined as the total percentage of participants whose best overall response (BOR) is either a complete response or partial response divided by the total percentage of participants who are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung (NSCL), and Gastric).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 58 months
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BMS-986148 Mesothelioma | BMS-986148+Nivolumab Mesothelioma | BMS-986148 Ovarian | BMS-986148+Nivolumab Ovarian | BMS-986148 Pancreatic | BMS-986148+Nivolumab Pancreatic | BMS-986148 NSCLC | BMS-986148+Nivolumab NSCLC | BMS-986148 Gastric | BMS-986148+Nivolumab Gastric
Number analyzed (Participants) | 25 | 13 | 22 | 2 | 18 | 6 | 4 | 2 | 3 | 1
Percentage of participants | 4.0 [0.1 to 20.4] | 23.1 [5.0 to 53.8] | 9.1 [1.1 to 29.2] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

11. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time between the date of first response and the subsequent date of objectively documented disease progression or death, whichever occurs first. Participants are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung (NSCL), and Gastric).
Time Frame: Up to 58 months
Population: Per-protocol, data for this Outcome Measure was collected by disease irrespective of dose. All response evaluable participants are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung Cancer (NSCLC), and Gastric).
Measure: Median (Full Range); unit: Months
Arm/Group | BMS-986148 Mesothelioma | BMS-986148+Nivolumab Mesothelioma | BMS-986148 Ovarian | BMS-986148+Nivolumab Ovarian | BMS-986148 Pancreatic | BMS-986148+Nivolumab Pancreatic | BMS-986148 NSCLC | BMS-986148+Nivolumab NSCLC | BMS-986148 Gastric | BMS-986148+Nivolumab Gastric
Number analyzed (Participants) | 1 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Months | 29.7 [29.7 to 29.7] | 8.97 [5.1 to 13.3] | NA [3.0 to 20.0] — Median not reached due to insufficient number of events |  |  |  |  |  |  |

12. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time from the first dose of study medication to the date of the first objective documentation of tumor progression or death due to any cause. Progression is defined with at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm. Participants who did not progress nor died will be censored on the date of their last tumor assessment. Participants are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung (NSCL), and Gastric).
Time Frame: Up to 58 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- BMS-986148 Pancreatic Part 1B: Part 1B Dose Escalation: BMS-986148 starting with a dose of 0.4 mg/kg IV QW to a dose of 0.6 mg/kg IV QW for 3 weeks and 1 week off in a 28-day cycle
- BMS-986148 Pancreatic: Part 1A Dose Escalation: BMS-986148 starting with a dose of 0.8 mg/kg IV Q3W to a dose of 1.6 mg/kg IV Q3W in a 21-day cycle
  Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
Arm/Group | BMS-986148 Mesothelioma | BMS-986148+Nivolumab Mesothelioma | BMS-986148 Ovarian | BMS-986148+Nivolumab Ovarian | BMS-986148 Pancreatic Part 1B | BMS-986148 Pancreatic | BMS-986148+Nivolumab Pancreatic | BMS-986148 NSCLC | BMS-986148+Nivolumab NSCLC | BMS-986148 Gastric | BMS-986148+Nivolumab Gastric
Number analyzed (Participants) | 25 | 13 | 22 | 2 | 7 | 11 | 6 | 4 | 2 | 3 | 1
Months | 2.56 [1.41 to 4.01] | 5.19 [2.56 to 12.06] | 2.79 [1.28 to 4.17] | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | 1.64 [1.45 to 1.71] | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | 1.66 [1.22 to 2.14] | 1.49 [1.15 to 5.65] | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate)

13. Secondary Outcome: Progression Free Survival Rate (PFSR) at Week t
Description: Progression free survival rate is defined as the proportion of participants who remain progression free and surviving at 't' weeks (t=4-12 months). The proportion will be calculated by the product-limit method (Kaplan-Meier estimate) which takes into account censored data. Participants are grouped by cohorts (Mesothelioma, Pancreatic, Ovarian, Non-smell Cell Lung (NSCL), and Gastric).
Time Frame: Total PFS assessed between 4 and 12 months, PFSR at months 4 and 6 to be reported
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | BMS-986148 Mesothelioma | BMS-986148+Nivolumab Mesothelioma | BMS-986148 Ovarian | BMS-986148+Nivolumab Ovarian | BMS-986148 Pancreatic Part 1B | BMS-986148 Pancreatic | BMS-986148+Nivolumab Pancreatic | BMS-986148 NSCLC | BMS-986148+Nivolumab NSCLC | BMS-986148 Gastric | BMS-986148+Nivolumab Gastric
Number analyzed (Participants) | 25 | 13 | 22 | 2 | 7 | 11 | 6 | 4 | 2 | 3 | 1
Proportion of participants
  4 months | 0.35 [0.15 to 0.54] | 0.65 [0.37 to 0.93] | 0.40 [0.18 to 0.62] | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate)
  6 months | 0.30 [0.11 to 0.49] | 0.47 [0.17 to 0.76] | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate) | NA [NA to NA] — Median, Lower Limit and Upper Limit are NA for Kaplan-Meier estimate because no observations were available for calculation of estimate (or confidence of estimate)

14. Secondary Outcome: Changes in QT Corrected by the Fridericia Formula (QTcF) From Baseline, at Selected Times
Description: Changes of participants in QT corrected by the fridericia formula (QTcF) Interval from baseline at <= 30 msec, >30 - <= 60 msec, and > 60 msec grouped by dose + dose regimen
Time Frame: Up to 58 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS 1.2MG/KG Q3W Ex | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab
Number analyzed (Participants) | 2 | 2 | 3 | 8 | 10 | 8 | 51 | 8 | 4 | 30
Participants
  <= 30 msec, | 1 | 2 | 2 | 6 | 9 | 8 | 37 | 5 | 3 | 23
  >30 - <= 60 msec | 1 | 0 | 1 | 2 | 1 | 0 | 12 | 3 | 1 | 7
  > 60 msec | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0

15. Secondary Outcome: Number of Participants With Anti-Drug Antibody (ADA)
Description: Number of participants with anti-drug antibody (ADA) status grouped by dose + dose regimen.
  Data was not collected for this outcome measure.
Time Frame: Up to 58 months
Population: All ADA evaluable participants
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W Es | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab | BMS 1.2MG/KG Q3W Ex
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to 100 days post last dose (Up to 6 months)
Groups:
- BMS-986148 1.2MG/KG Q3W: Part 1A Dose Escalation BMS-986148 1.2 mg/kg IV Q3W
  Part 2 Dose Expansion: BMS-986148 1.2 mg/kg IV Q3W restricted to five tumor types: 1) mesothelioma; 2) pancreatic; 3) ovarian; 4) NSCLC; and 5) gastric cancer
Arm/Group | BMS-986148 0.1MG/KG Q3W | BMS-986148 0.2MG/KG Q3W | BMS-986148 0.4MG/KG Q3W | BMS-986148 0.8MG/KG Q3W | BMS-986148 1.6MG/KG Q3W | BMS-986148 1.2MG/KG Q3W | BMS-986148 0.4MG/KG QW | BMS-986148 0.6MG/KG QW | BMS-986148 0.8MG/KG Q3W+Nivolumab
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/2 | 3/3 | 5/8 | 7/10 | 38/59 | 7/8 | 4/4 | 22/30
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 1/3 | 5/8 | 4/10 | 32/59 | 6/8 | 3/4 | 21/30
Other Adverse Events (participants affected / at risk) | 1/2 | 2/2 | 3/3 | 8/8 | 10/10 | 57/59 | 8/8 | 4/4 | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986148 0.1MG/KG Q3W (N=2) | BMS-986148 0.2MG/KG Q3W (N=2) | BMS-986148 0.4MG/KG Q3W (N=3) | BMS-986148 0.8MG/KG Q3W (N=8) | BMS-986148 1.6MG/KG Q3W (N=10) | BMS-986148 1.2MG/KG Q3W (N=59) | BMS-986148 0.4MG/KG QW (N=8) | BMS-986148 0.6MG/KG QW (N=4) | BMS-986148 0.8MG/KG Q3W+Nivolumab (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Duodenal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 4
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 13 | 2 | 2 | 8
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS-986148 0.1MG/KG Q3W (N=2) | BMS-986148 0.2MG/KG Q3W (N=2) | BMS-986148 0.4MG/KG Q3W (N=3) | BMS-986148 0.8MG/KG Q3W (N=8) | BMS-986148 1.6MG/KG Q3W (N=10) | BMS-986148 1.2MG/KG Q3W (N=59) | BMS-986148 0.4MG/KG QW (N=8) | BMS-986148 0.6MG/KG QW (N=4) | BMS-986148 0.8MG/KG Q3W+Nivolumab (N=30)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 2 | 1 | 2
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 5 | 0 | 0 | 2
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 3
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 1 | 4 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 3 | 15 | 4 | 1 | 5
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 3 | 5 | 0 | 0 | 6
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 16 | 3 | 1 | 10
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 8 | 13 | 1 | 1 | 5
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 5 | 1 | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 5 | 0 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 5 | 7 | 30 | 3 | 1 | 13
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 1
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 4 | 4 | 17 | 0 | 1 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 10 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Early satiety (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 5 | 8 | 32 | 3 | 3 | 15
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 5 | 3 | 1 | 5
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 2 | 8 | 0 | 0 | 2
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 3 | 14 | 1 | 2 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 6 | 33 | 3 | 3 | 10
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 3 | 5 | 35 | 2 | 3 | 12
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 5 | 18 | 2 | 2 | 5
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 8 | 2 | 2 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Blood sodium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 3 | 0 | 4 | 0 | 0 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 1 | 6 | 5 | 26 | 2 | 2 | 11
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 3 | 0 | 4 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 2 | 4 | 0 | 1 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2 | 1 | 10 | 1 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 5 | 0 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 4
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 7 | 1 | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 3 | 5 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 6 | 1 | 2 | 4
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 3 | 6 | 0 | 1 | 4
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 0 | 4 | 1 | 0 | 6
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 2 | 13 | 0 | 0 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 5 | 19 | 1 | 1 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 3 | 7 | 2 | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 7 | 1 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-11-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT02341625/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT02341625/SAP_001.pdf